CLINICAL TRIAL: NCT01661348
Title: Reduction of Post Operative Wound Complications in Patients Undergoing Cesarean Delivery With the Use of the Prevena Incision Management System
Brief Title: The Use of the Prevena Incision Management System to Reduce Post-operative Cesarean Delivery Wound Complications
Status: Withdrawn | Type: Observational
Why Stopped: Did not receive funding.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: Prevena-Smith
Record Dates: First submitted 2012-07-26; First posted 2012-08-09 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Pregnancy
Keywords: Cesarian section; Pregnancy; Incision management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prevena System placement: Subjects randomized to this group will receive standard skin preparation and closure followed by application of Prevena Incision Management System (Kinetic Concepts, Inc; San Antonio, TX) negative pressure wound therapy unit (experimental group).
- Standard of care postoperative care: Subjects randomized to this group will receive a standard surgical skin preparation, closure, and dressing (control group).

SUMMARY:
Aim 1: Assess the effectiveness of the Prevena Incision Management System in decreasing postoperative surgical site infections in the obese parturient undergoing non-emergent cesarean delivery.

Aim 2: Assess patient satisfaction after using the Prevena Incision Management System following a non-emergent cesarean delivery.

Our overall long term goal is to reduce morbidity and incidence of surgical site infection (SSI) in obese parturient who undergo non-emergent cesarean delivery.

DETAILED DESCRIPTION:
In the United States, the cesarean delivery rate continues to rise. In 2007, approximately 32% of all births occurred by Cesarean delivery, translating to 1.4 million women who underwent this operative procedure. Oklahoma is on par with the national average, with 33.6 % of births occuring by Cesarean delivery (1). Although in 2006 Cesarean delivery was the most commonly performed surgical procedure in the United States, it remains vulnerable to common, as well as rare, complications. Despite continued advances in surgical and aseptic technique, surgical site infections (SSI) continue to be an area of concern for patients, physicians, hospitals, and insurers.

In addition to their negative impact on patient quality of life, surgical site infections (SSI) have been estimated to require an additional three thousand dollars per infection in healthcare expenditure (2). In the surgical patient, it has been estimated that SSI account for 25 to 38% of hospital acquired infections (3-4) and 2-5% of patients undergoing surgery of any type will develop a SSI (5). In cesarean delivery in particular, rates of SSI are between 3 to 15%, depending on the population, definition of SSI, and modifiable risk factors (6). In particular, one factor shown to increase risk of SSI in multiple studies is obesity with odds ratios 1.1-4.79 depending on degree of BMI stratification (6-8). Given its prevalence and cost, SSI represents a postoperative complication with far reaching consequences and making it an area of increasing focus for research.

Recently, negative pressure wound therapy has come to the forefront in demonstrating improved healing and reduced complications in open and closed surgical wounds of various types. A review of the literature illustrates that prophylactic negative pressure wound therapy device effectiveness in reducing SSI has not been widely evaluated in cesarean deliveries. The goal of this study is to evaluate wound infection rates with the use of the Prevena Incision Management System in obese patients undergoing non-emergent cesarean delivery at a tertiary care center. We propose to initiate a randomized clinical trial of the Prevena Incision Management System in a novel population of patients at high risk of surgical site infection. Given the possibility of unexpected challenges, we propose to begin this project with a pilot study in order to help elucidate factors that may need to be including in a larger study in the future. Also, we anticipate that the pilot study will give us a better insight into the rates of wound complications and potential difference between groups in order to better power a larger study.

Rationale for study: Obese patients undergoing Cesarean deliveries have frequent SSIs secondary to modifiable and non-modifiable risk factors. A randomized controlled trial of Prevena Incision Management System, a single use negative pressure therapy unit designed for placement over clean closed surgical incisions, will help reduce rates of surgical site infections and increase the overall quality of life of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than or equal to 18-years-of-age having a non-emergent Cesarean delivery, primary or repeat procedure, without evidence of active infection at the time of the procedure

  * Patient with BMI ≥ 30 kg/m2 at the time of hospital admission
  * Patient able to provide informed consent for study
  * Patient able to complete follow-up

Exclusion Criteria:

* Males

  * Females under the age of 18
  * Known sensitivity to silver due to the presence of silver in the skin interface layer of the Prevena
  * Patients unable to consent
  * Patients in active labor
  * Patients with a diagnosis of preterm premature rupture of membranes
  * Patients with known or suspected infection at the time of Cesarean delivery
  * Patients with a contraindication to use of the Prevena Incision Management System

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All eligible patients will be approached for consent to participate in the study prior to surgical procedure.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Wound Infections | The percent of patients with wound infections will be summarized at the 5-7 day post-operative assessment, the 14-21 day post-operative assessment, and the 6-week follow-up visit. The rate of wound infections will be evaluated at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Smith, MD, Principal Investigator — University of Oklahoma; Elise Eckhardt, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States